CLINICAL TRIAL: NCT06932328
Title: A Randomized, Double-Blind, Dose-Exploration, Multicenter Phase II Clinical Trial to Evaluate the Efficacy and Safety of Qin Qiao Yan Shu Granules in the Treatment of Acute Pharyngitis (Exterior Wind-Heat Syndrome)
Brief Title: Qinqiao Yan Shu Granules for the Treatment of Acute Pharyngitis (Exterior Wind-Heat Syndrome) Phase II Clinical Trial
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jianmin Pharmaceutical Group Co., LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: JM-2024-04
Record Dates: First submitted 2025-04-10; First posted 2025-04-17 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Acute Pharyngitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Qinqiao Yanshu Granules High - dose group (Experimental)
  Interventions: Drug: Qinqiao Yanshu Granules
- Qinqiao Yanshu Granules Low - dose group (Experimental)
  Interventions: Drug: Qinqiao Yanshu Granules
- Qinqiao Yanshu Granules Extremely low - dose group (Experimental)
  Interventions: Drug: Qinqiao Yanshu Granules

INTERVENTIONS:
Drug: Qinqiao Yanshu Granules — High - dose group: Dissolve in boiling water and take 1 bag each time, 3 times a day, half an hour before meals; Low - dose group: Dissolve in boiling water and take 1 bag each time, 3 times a day, half an hour before meals; Extremely low - dose group: Dissolve in boiling water and take 1 bag each time, 3 times a day, half an hour before meals; Rescue medication: Paracetamol tablets. During the trial, if the subject's body temperature exceeds 38.5°C (including 38.5°C), rescue medication can be added. Use it according to the instructions and doctor's advice and record it truthfully.

SUMMARY:
Trial Objectives and Exploration Indicators：

1. To explore the improvement effect of different doses of Qinqiao Yanshu Granules on the symptoms/conditions and TCM syndromes of acute pharyngitis (Wind - Heat Exogenous Syndrome), and its effect on shortening the course of the disease.
2. To observe the safety of the clinical application of Qinqiao Yanshu Granules. Overall Trial Design：A block - randomized, double - blind, dose - escalation, multicenter clinical trial design was adopted.

Sample Size：It is planned to enroll 72 cases in each group (high - dose group, low - dose group, and extremely low - dose group), with a total of 216 cases.

Investigational Products：Experimental groups:

1. High - dose group: Specification: 12g/bag;
2. Low - dose group: Specification: 12g/bag.

Control group:

(1) Extremely low - dose group: Specification: 12g/bag.

Rescue medication:

(1) Paracetamol tablets: Specification: 0.5g/tablet. Dosage and Administration： High - dose group: Dissolve in boiling water and take 1 bag each time, 3 times a day, half an hour before meals; Low - dose group: Dissolve in boiling water and take 1 bag each time, 3 times a day, half an hour before meals; Extremely low - dose group: Dissolve in boiling water and take 1 bag each time, 3 times a day, half an hour before meals; Rescue medication: Paracetamol tablets. During the trial, if the subject's body temperature exceeds 38.5°C (including 38.5°C), rescue medication can be added. Use it according to the instructions and doctor's advice and record it truthfully.

Treatment Course：5 days Efficacy Indicators：

1) The disappearance rate of pharyngeal pain 3 days and 5 days after treatment; 2) The change value of the pharyngeal pain VAS score compared with the baseline 5 days after treatment; 3) The time to disappearance of pharyngeal pain; 4) The effective rate of pharyngeal signs 5 days after treatment; 5) The clinical cure rate of the disease 5 days after treatment; 6) The efficacy of TCM syndromes 5 days after treatment; 7) The disappearance rate of single symptoms 5 days after treatment; 8) The frequency of rescue drug use. Measurement and Definition of Endpoint Indicators：

1. The criterion for the disappearance of pharyngeal pain: The pharyngeal pain VAS score drops to 0 points and persists for 24 hours or more.
2. Pharyngeal pain VAS score:

   Starting from the evaluation time of the VAS score during the screening period, the subject evaluates once every 24 hours (±1 hour) and records the most severe degree of pharyngeal pain in the past 24 hours in the diary card.
3. The criterion for the effective rate of pharyngeal signs: "Effective" is defined as a decrease of at least 1 point in the pharyngeal sign score. The effective rate = (Number of effective cases / Total number of cases) × 100%.
4. The criterion for the clinical cure of the disease: The clinical symptoms of the disease disappear, and the pharyngeal signs are reduced to mild or less. The cure rate = (Number of cured cases / Total number of cases) × 100%.
5. The definition of the efficacy of TCM syndromes:

Efficacy of TCM syndromes: Cure means that the TCM syndrome score decreases by ≥ 95%; Marked effect means that the TCM syndrome score decreases by ≥ 70% and < 95%; Effective means that the TCM syndrome score decreases by ≥ 30% and < 70%; Ineffective means that it does not meet the above criteria.

The change value of the pharyngeal pain VAS score compared with the baseline = The baseline pharyngeal pain VAS score - The pharyngeal pain VAS score on the 6th day.

Study Population；

Inclusion criteria:

1. Meeting the Western medical diagnostic criteria for acute pharyngitis;
2. Meeting the TCM syndrome differentiation criteria for Wind - Heat Exogenous Syndrome;
3. The course of the disease at the time of consultation ≤ 48 hours;
4. The pharyngeal pain VAS score ≥ 4 points and the pharyngeal sign score ≥ 1 point;
5. Aged between 18 and 65 years old (including the boundary values), regardless of gender;
6. Voluntarily participating in this clinical trial and signing the informed consent form.

Exclusion criteria:

1. Those with pharyngeal symptoms or inflammation caused by measles, scarlet fever, agranulocytosis, infectious mononucleosis, influenza, diphtheria, acute epiglottitis, acute carotid arteritis, etc.;
2. Those with concurrent acute sinusitis, acute laryngitis, suppurative tonsillitis, bronchitis, pneumonia;
3. Those with a modified Centor score ≥ 2, a body temperature peak > 38.5°C (axillary temperature) within 24 hours before this visit, a white blood cell count > 1.2 × ULN, a neutrophil percentage > 1.2 × ULN, and considered to be bacterial infections by the researcher;
4. Those with concurrent severe primary diseases of the cardiovascular and cerebrovascular system, liver, kidney, hematopoietic system, endocrine system, and mental diseases;
5. Those with a history of thyroid - related diseases such as hyperthyroidism and hypothyroidism;
6. Those with laboratory test results

ELIGIBILITY:
Inclusion Criteria:

1. Meeting the Western medicine diagnostic criteria for acute pharyngitis.
2. Meeting the TCM syndrome differentiation criteria for the syndrome of wind-heat invading the exterior.
3. The disease course at the time of visit is ≤ 48 hours.
4. The VAS score for pharyngeal pain is ≥ 4 points, and the pharyngeal sign score is ≥ 1 point.
5. Age between 18 and 65 years old (including the boundary values), regardless of gender.
6. Voluntarily participating in this clinical trial and signing the informed consent form.

Exclusion Criteria:

1. Those with pharyngeal symptoms or inflammation caused by measles, scarlet fever, agranulocytosis, infectious mononucleosis, influenza, diphtheria, acute epiglottitis, acute carotid arteritis, etc.
2. Those with concurrent acute sinusitis, acute laryngitis, suppurative tonsillitis, bronchitis, pneumonia.
3. Those with a modified Centor score ≥ 2 points, a peak body temperature > 38.5°C (axillary temperature) within 24 hours before this visit, a white blood cell count > 1.2 × ULN, a neutrophil percentage > 1.2 × ULN, and suspected bacterial infection considered by the researcher.
4. Those with concurrent severe primary diseases of the cardiovascular and cerebrovascular system, liver, kidney, hematopoietic system, endocrine system, and mental diseases.
5. Those with a history of thyroid-related diseases such as hyperthyroidism or hypothyroidism.
6. Those with laboratory test results indicating ALT > 1.2 × ULN, AST > 1.2 × ULN, or Cr > 1 × ULN. Any one of these conditions will lead to exclusion.
7. Those who have used any other drugs for the treatment of acute pharyngitis, including drugs for relieving pharyngeal pain (such as traditional Chinese medicines, glucocorticoids, non-steroidal anti-inflammatory drugs, etc.) within 48 hours before this visit.
8. Those who are allergic to the ingredients or excipients of the test drug.
9. Pregnant or lactating women.
10. Those suspected of or with a confirmed history of alcohol or drug abuse.
11. Patients who have participated in or are currently participating in other clinical trials within the past month.
12. Patients considered by the researcher to be unsuitable for participating in this clinical trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2025-03-26 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The disappearance rate of pharyngeal pain 3 and 5 days after treatment | 3days/5days

CONTACTS AND LOCATIONS:
Locations (7):
- China (7):
  - The First Affiliated Hospital of Heilongjiang University of Chinese Medicine, Harbin, Heilongjiang
  - The First Affiliated Hospital of Hunan University of Chinese Medicine, Changsha, Hunan
  - Affiliated Hospital of Changchun University of Chinese Medicine, Changchun, Jilin
  - Affiliated Hospital of Shandong University of Traditional Chinese Medicine, Jinan, Shandong
  - The Affiliated Traditional Chinese Medicine Hospital of Southwest Medical University, Luzhou, Sichuan
  - First Affiliated Hospital of Tianjin University of Traditional Chinese Medicine, Tianjin, Tianjin Municipality
  - Wenzhou Hospital of Traditional Chinese Medicine, Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided